CLINICAL TRIAL: NCT06513650
Title: Mechanism-based Therapy of Hypotensive Syncope
Acronym: 2STEPtherapy
Status: Recruiting | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 09C408
Record Dates: First submitted 2024-07-16; First posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Syncope, Vasovagal, Neurally-Mediated
MeSH Terms: conditions — Syncope, Vasovagal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Drug deprescring and drug addition: This multicentre, prospective, observational, pragmatic study on long-term therapy of hypotensive syncope consists of two distinct twin substudies to be undergone in parallel:
  1. the Drug-deprescribing substudy wants to assess a strategy aimed to increase BP by deprescribing of hypotensive drugs in hypertensive patients affected by drug-related syncope, and;
  2. the Drug-addition substudy wants to assess a therapeutic strategy aimed at increasing BP with fludrocortisone in syncopal patients with drug-unrelated permanent or intermittent hypotension.

SUMMARY:
The aim of this study is to assess the efficacy of a therapeutic strategy aimed to increase 24-hour systolic blood pressure (SBP) values, assessed by 24-hour ambulatory blood pressure monitoring (ABPM), in reducing syncope recurrences in patients affected by hypotensive syncope during one year of follow-up.

DETAILED DESCRIPTION:
This multicentre, prospective, observational, pragmatic study on long-term therapy of hypotensive syncope consists of two distinct twin substudies to be undergone in parallel:

1. the Drug-deprescribing substudy wants to assess a strategy aimed to increase BP by deprescribing of hypotensive drugs in hypertensive patients affected by drug-related syncope, and;
2. the Drug-addition substudy wants to assess a therapeutic strategy aimed at increasing BP with fludrocortisone in syncopal patients with drug-unrelated permanent or intermittent hypotension.

Inclusion criteria

1. Patients >18-year-old with a clinical diagnosis of severe, recurrent reflex syncope, refractory to education and life-style measures (according to the criteria of ESC guidelines) AND a diagnosis of hypotensive syncope defined as:

   * Persistent or intermittent hypotension during 24-hour ABPM (ABPM1) AND/OR
   * Reproduction of syncope during the Short Cardiovascular Autonomic Function Assessment (SCAFA) that consists in carotid sinus massage (CSM), 3-min active stand test, and head-up tilt test (TT) performed one after another in an uninterrupted sequence as a single procedure in a tilt table.
2. Clinical indication to deprescribing of antihypertensive drugs or to prescribing of fludrocortisone therapy, as appropriate, according to the clinical practice of the investigator Exclusion criteria

1. Age <18 years 2. Cardioinhibitory reflex syncope during SCAFA tests 3. Competing causes of syncope 4. Severe cardiac disease, previous stroke or transient ischaemic attack. 5. Patients who refused drug therapy 6. Non-severe forms of syncope, i.e., patients with rare and mild episodes occurring in low-risk situations in the presence of distinct and preventable triggers.

7. Contraindication to fludrocortisone Therapy The strategy of deprescribing (withdrawal or dose reduction) is empirically based on the usual clinical practice of the investigators and is targeted to achieve an absolute value ≥134 mmHg and/or an increase ≥12 mmHg of 24-hour SBP.

The initial recommended dose of fludrocortisone is 0.2 md/day, accepted range is 0.1 to 0.3 mg and is targeted to achieve an absolute value of ≥116 mmHg and/or an increase of ≥9 mmHg of 24-hour SBP.

30-day optimization period A period up to 30 days is allowed to optimize therapy, if necessary, with the goal to achieve the above targets of mean 24-hour SBP during an ABPM performed at the end of this period (ABPM2). Subsequent follow-up visits are performed at 4, 8 and 12 months.

Primary endpoints

* The primary endpoint of the Drug-deprescribing subgroup is the comparison of syncopal recurrences (time to first recurrence and syncope burden) at one year in patients who achieved a mean absolute value of ≥134 mmHg and/or an increase ≥12 mmHg of 24-hour SBP on ABPM2 (Target) with those of patients who did not (No target).
* The primary endpoint of the Drug-addition subgroup is the comparison of syncopal recurrences (time to first recurrence and syncope burden) at one year in patients who achieved a mean absolute value of ≥116 mmHg and an increase of ≥9 mmHg of 24-hour SBP on ABPM2 (Target) with those of patients who did not (No target).

Secondary endpoints

* Comparison between the burden of syncope and presyncope during the year before with that during the year after enrolment
* Exploratory analyses with the aim to identify eventual different targets that are better predictor of efficacy of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18-year-old with a clinical diagnosis of severe, recurrent reflex syncope, refractory to education and life-style measures (according to the criteria of ESC guidelines) AND a diagnosis of hypotensive syncope defined as:
* Persistent or intermittent hypotension during 24-hour ABPM (ABPM1) AND/OR
* Reproduction of syncope during the Short Cardiovascular Autonomic Function Assessment (SCAFA) that consists in carotid sinus massage (CSM), 3-min active stand test, and head-up tilt test (TT) performed one after another in an uninterrupted sequence as a single procedure in a tilt table.

  2. Clinical indication to deprescribing of antihypertensive drugs or to prescribing of fludrocortisone therapy, as appropriate, according to the clinical practice of the investigator

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Age <18 years
  2. Cardioinhibitory reflex syncope during SCAFA tests
  3. Competing causes of syncope
  4. Severe cardiac disease, previous stroke or transient ischaemic attack.
  5. Patients who refused drug therapy
  6. Non-severe forms of syncope, i.e., patients with rare and mild episodes occurring in low-risk situations in the presence of distinct and preventable triggers.
  7. Contraindication to fludrocortisone
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Time to first syncope recurrenceSyncope | 4 months
  • The primary endpoint of the Drug-deprescribing subgroup is the comparison of syncopal recurrences (time to first recurrence and syncope burden) at one year in patients who achieved a mean absolute value of ≥134 mmHg and/or an increase ≥12 mmHg of 24-hour SBP on ABPM2 (Target) with those of patients who did not (No target). • The primary endpoint of the Drug-addition subgroup is the comparison of syncopal recurrences (time to first recurrence and syncope burden) at one year in patients who achieved a mean absolute value of ≥116 mmHg and an increase of ≥9 mmHg of 24-hour SBP on ABPM2 (Target) with those of patients who did not (No target).

CONTACTS AND LOCATIONS:
Locations (8):
- University of marseille Aix en Provence, Marseille, France
- Italy (4):
  - IRCCS Istituto Auxologico Italiano, Milan, MI
  - University of Florence, Florence
  - ospdali del Tigullio, Lavagna
  - Università della Campania Vamvitelli, Naples
- AMC Universisty of Amsterdam, Amsterdam, Netherlands
- University of Barcelona Vall d'Ebron, Barcelona, Spain
- Karolinska Institut, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No